CLINICAL TRIAL: NCT04856826
Title: Placement of Peripheral Venous Catheters Under Echo Guidance in a Post-emergency Medical Service
Acronym: KatECHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC19.419
Record Dates: First submitted 2021-01-11; First posted 2021-04-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Catheterization, Peripheral; Echography; Hospital Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- echo guidance (Experimental): insertion of a peripheral venous catheter with ultrasound guidance and therapeutic communication
  Interventions: Device: ultrasound guidance and therapeutic communication
- conventional (No Intervention): insertion of a peripheral venous catheter conventionally

INTERVENTIONS:
Device: ultrasound guidance and therapeutic communication — insertion of a peripheral venous catheter with ultrasound guidance and therapeutic communication
  Arms: echo guidance

SUMMARY:
Compare the number of attempts to place a peripheral venous catheter in the group of patients hospitalized in the post-emergency unit and benefiting from echo guidance and therapeutic communication, to the group of patients hospitalized on the post-emergency unit using traditional technique.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the post-emergency unit
* Requiring the placement of a venous catheter in the post-emergency unit
* Affiliation to social security or benefiting from such a scheme
* Informed and written consent signed

Exclusion Criteria:

* Protected person (art. L1121-5 to L1121-8 of the CSP)
* Patient included in another interventional study
* Patient already included for a first catheter placement in the post-emergency unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
successful placement of a venous catheter on the first attempt | within the hour after insertion of peripheral venous catheter
  percentage of successful placement of a venous catheter on the first attempt

SECONDARY OUTCOMES:
patient experience | within the hour after insertion of peripheral venous catheter
  not validated Satisfaction questionnaire and pain scale. score between 0 and 30 corresponding to high satisfaction
number of attempts to insert a peripheral venous catheter | within the hour during insertion of peripheral venous catheter
  Average in each group of the number of attempts
number of calls for a second nurse in the service | within the hour during insertion of peripheral venous catheter
  Average in each group of the number of service's interveners for a catheter placement
number of calls to a nurse anesthetist | within the hour during insertion of peripheral venous catheter
  Average in each group of the number of external interveners
location of the final placement site | within the hour during insertion of peripheral venous catheter
  Proportion of patients in each group according to the location of the final placement site
the caliber of the catheter placed | within the hour during insertion of peripheral venous catheter
  Proportion of patients in each group according to the caliber of the catheter placed
infectious or thromboembolic events | 4 days
  total number of infectious or thromboembolic events at the implantation site during the patient's stay in the post-emergency unit
duration of catheter placement | within the hour during insertion of peripheral venous catheter
  Average duration, in minutes, of catheter placement in each group
functional life of the catheter | 4 days
  functional life of the catheter, by group.
Satisfaction of nursing staff | at the end of study inclusion, at 6 month
  not validated Satisfaction questionnaire for nursing staff in the post-emergency unit . score between 0 and 55 corresponding to a high satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Perrine Dumanoir, Study Chair — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736